CLINICAL TRIAL: NCT01152762
Title: Effectiveness of Standardized Respiratory Physiotherapy in Primary Care in Patients With Mild COPD and Its Economic Assessment
Brief Title: Effectiveness of Standardized Respiratory Physiotherapy in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Maria Montserrat Ingles Novell, Jordi Gol i Gurina Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07/42
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: COPD
Keywords: Physiotherapy, COPD, effectiveness, primary care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standardized Respiratory Physiotherapy (Experimental): Standardized Respiratory Physiotherapy is the intervention in all selected patients
  Interventions: Procedure: Standardized Respiratory Physiotherapy

INTERVENTIONS:
Procedure: Standardized Respiratory Physiotherapy — Standardized Respiratory Physiotherapy during 6 months

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a very important public health problem and one of the most common lung diseases in the world, with repercussions on mortality and high economic costs. The World Health Organization estimates that COPD is the fifth most common disease in the world and the fourth leading cause of death. It is expected to grow in prevalence and mortality over the coming decades; it is estimated that in 2020, it will be the third most common cause of death worldwide.

Primary care is the main ambit in the management of these patients, in fact, it is where most patients with COPD are visited. However, a high proportion of these patients only receive chest physiotherapy treatment in hospitals, and the implementation of this kind of treatment in primary care is still very uncommon.

Hypothesis: There is effectiveness on the quality of life and various predictive factors of mortality (BODE index, six-minute walk distance, FEV1, dyspnea, and body mass index) and the economic impact of a Standardized Respiratory Physiotherapy program conducted in Primary Care (FREAP) in patients with moderate COPD at 6 months after its implementation.

DETAILED DESCRIPTION:
AIMS

To evaluate the effectiveness on the quality of life and various predictive factors of mortality (BODE index, six-minute walk distance, FEV1, dyspnea, and body mass index) and the economic impact of a Standardized Respiratory Physiotherapy program conducted in Primary Care (FREAP) in patients with moderate COPD at 6 months after its implementation.

METHOD

Design: Randomized controlled trial

Location: Tarragona-Reus Primary Care Area of the Catalan Health Service. 14 primary care centres were involved in the project (8 from the Reus-Altebrat Primary Care Service and 6 from the Tarragona-Valls Primary Care Service) and 8 units of physiotherapy.

Participants: 129 patients with moderate COPD treated by primary care teams.

Intervention: FREAP program for 6 months. It consisted of an initial health education session conducted in the primary care health centre, three sessions a week for three weeks of breathing exercises and aerobic, physical training in the primary care health centre and a monthly monitoring appointment for the breathing exercises and training for five months in the patient's home. Altogether, 10 sessions in the primary care health center and 5 sessions at the patients' house. Patients randomized in the control group continued with their usual clinical practice.

Main effect measures: Quality of life (St. George Respiratory Questionnaire -SGRQ-). Predictive factors of mortality (BODE index, six-minute walk distance, FEV1, dyspnea, and body mass index). Economic cost of implementing the FREAP program.

ELIGIBILITY:
Inclusion Criteria:

* Mild COPD diagnostic by GOLD criteria.
* Absence of contraindications for walk tests and training.
* Disponibility.
* Age between 40 and 74 years old.

Exclusion Criteria:

* Patients with treatment of oxygen or domiciliary oxygen therapy.
* Communication deficience(dementia, terminal illness, illiteracy).
* Informed consent not available.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire | Six months
  Quality of life Questionnaire

SECONDARY OUTCOMES:
BODE index | Six months
  Is a complex index that measures dyspnea, FEV1, BMI, and six-minute walk distance

CONTACTS AND LOCATIONS:
Overall Officials: Maria Montserrat Ingles Novell, Principal Investigator — Catalan Institute of Health
Locations (1):
- Catalan Health Institute, Reus, Tarragona, Spain